CLINICAL TRIAL: NCT01450657
Title: Observational Clinical Trials of Kibow Biotics (a Patented and Proprietary Probiotic Dietary Supplement) in Chronic Kidney Failure Patients, in Conjunction With Standardized Care of Treatment
Brief Title: Observational Study of Kibow Biotics in Chronic Kidney Failure Patients
Status: Completed | Type: Observational
Sponsor: Kibow Pharma (Industry)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: KIB002
Record Dates: First submitted 2011-09-26; First posted 2011-10-12 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Chronic Kidney Failure
Keywords: Chronic Kidney failure stage three and four; Probiotics; Kibow Biotics; Dialysis; Gut based uremic toxin removal
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic Kidney Failure 3/4
  Interventions: Dietary Supplement: Kibow Biotics/Renadyl

INTERVENTIONS:
Dietary Supplement: Kibow Biotics/Renadyl — Month 1, one capsule three times daily (90 colony forming units); Month 2, two capsules three times daily (180 CFU's); Month 3 & 4, three capsules three times daily (270 CFU's). Months 5 & 6 are washout periods, in which the patient receives no product. All parameters are still monitored by the study site during months 5 & 6. All medical, physical, clinical, QOL and other parameters will be monitored as well.
  Other Names: Kibow Biotics

SUMMARY:
A specifically formulated probiotic product comprised of defined and tested microbial strains may afford renoprotection in what has been generally called "Enteric DialysisTM". However, it is also referred to as enteric toxin reduction technology. Our hypothesis is to assess the potential benefits in devising a bowel-based probiotic formulation (Kibow® Biotics/RenadylTM) as a dietary supplement product for patients undergoing standardized care of treatment for their CKD stage 3 and stage 4 conditions.

DETAILED DESCRIPTION:
Probiotics are increasingly utilized clinically. As their safety and health benefits are established, it is reasonable to anticipate that probiotic bacteria will be incorporated into a growing number of clinical regimens, as a dietary supplement.

Extensive in vitro R&D investigations in Kibow's laboratories

Bacterial strains studied were a mixture of patented and proprietary strains of Streptococcus thermophilus (KB27), Lactobacillus acidophilus (KB31) and Bifidobacterium longum (KB35).

Oral administration of these bacterial formulations, tested in the 5/6th nephrectomized rat model (at Thomas Jefferson University, Phila., PA) and minipig model (at Indiana University, Indianapolis, IN), decreased both blood urea nitrogen (BUN) and serum creatinine (Scr) levels.

Two independent veterinarians investigated the effect of Kibow Biotics® in cats and dogs (of both genders and varying body weights) with moderate to severe kidney failure. Based on positive results, this formulation, marketed and distributed as AzodylTM, is currently licensed for veterinary applications to Vetoquinol USA.

Pilot scale studies, double blind, placebo controlled, cross-over studies for six months conducted in 45 patients in USA, Canada, Argentina, and Nigeria demonstrates reduction of BUN (P>95%) and improved quality of life (P>95%). Decrease in creatinine and uric acid levels were also observed. However, these studies were based on correlating the age of geriatric cats and dogs with moderate to significant kidney failure to human geriatric conditions. The proposed current study is being reevaluated based on correlating the weight basis of animal to human conditions. Hence, this is a does escalation study on ingestion of 1x (90 billion CFU/day), 2x (180 billion CFU/day), and 3x (270 billion CFU/day) dosages.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* CKD Stages 3 and 4 as documented by prior medical history
* Serum Creatinine >2.5 mg/dL
* Stable and on CKD status 3 and 4 at least for a year or more

Exclusion Criteria:

* Pregnant or nursing women
* Refusal to sign the informed consent form
* Documented to have HIV/AIDS/Liver disease
* Active dependency on drugs or alcohol
* Any non-related medical, debilitating disease/disorder that would interfere with adherence to this study
* Currently on anticoagulant therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient hospital setting.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
15-20% Changes in BUN. | Baseline, 1 month, 2 months, 3 months, 4 months, 6 months.
15-20% Change in Creatinine | Baseline, 1 month, 2 months, 3 months, 4 months, 6 months

SECONDARY OUTCOMES:
Quality of life outcome based on questionnaire. | Baseline, 1 month, 2 months, 3 months, 4 months, 6 months
To observe inflammatory and oxidative stress biomarkers. | Baseline, 1 month, 2 months, 3 months, 4 months, 6 months
  Observe inflammatory and stress markers in metabolites from blood serum.
Observation and analysis of patient fecal matter. | Baseline, 1 month, 2 months, 3 months, 4 months, 6 months
  Observation and analysis of patient fecal matter to determine bacterial flora levels that are present in the stool.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie DeLoach, M.D., Principal Investigator — Thomas Jefferson University, Philadelphia, PA
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Ranganathan N, Friedman EA, Tam P, Rao V, Ranganathan P, Dheer R. Probiotic dietary supplementation in patients with stage 3 and 4 chronic kidney disease: a 6-month pilot scale trial in Canada. Curr Med Res Opin. 2009 Aug;25(8):1919-30. doi: 10.1185/03007990903069249. PMID 19558344
- [Result] Ranganathan N, Ranganathan P, Friedman EA, Joseph A, Delano B, Goldfarb DS, Tam P, Rao AV, Anteyi E, Musso CG. Pilot study of probiotic dietary supplementation for promoting healthy kidney function in patients with chronic kidney disease. Adv Ther. 2010 Sep;27(9):634-47. doi: 10.1007/s12325-010-0059-9. Epub 2010 Aug 16. PMID 20721651